CLINICAL TRIAL: NCT02471157
Title: The Association of Hypogonadism and Post-operative Outcomes of Oncologic Surgery
Brief Title: Hormonal Predictors of Oncologic Surgery
Acronym: HPOS
Status: Completed | Type: Observational
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Other Study IDs: 1408015434
Record Dates: First submitted 2015-05-04; First posted 2015-06-15 (Estimated); Last update posted 2019-01-25 (Actual); Status verified 2019-01

CONDITIONS: Hypogonadism
MeSH Terms: conditions — Hypogonadism | interventions — Observation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Eugonadal: Eugonadal men
  Interventions: Other: Observation
- Hypogonadal: Hypogonadal men
  Interventions: Other: Observation

INTERVENTIONS:
Other: Observation

SUMMARY:
An observational trial to determine whether preoperative hormonal status predicts outcomes of oncologic surgery.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing above surgery for cancer

Exclusion Criteria:

* Started hormonal replacement in past two months

Min Age: 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Men undergoing renal, bladder, and colorectal surgery for cancer
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2015-01; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Length of Stay | 6 days, on average
  Length of post-operative stay
Complication rate, post-operative | 6 days, on average
  Complication rate during initial postoperative period
Complication rate, 30 day | 30 days
  Complication rate during the initial 30 days after surgery
Complication rate, 90 days | 90 days
  Complication rate during the initial 90 days after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Douglas Scherr, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medical College, New York, New York, United States